CLINICAL TRIAL: NCT02446626
Title: Xenodiagnosis After Antibiotic Treatment for Lyme Disease - Phase II Study
Brief Title: Xenodiagnosis After Antibiotic Treatment for Lyme Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Stony Brook University (Other); Mansfield Family Practice LLC (Other); Tufts Medical Center (Other); New York Medical College (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 150131; 15-I-0131
Record Dates: First submitted 2015-05-13; First posted 2015-05-18 (Estimated); Results first posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2022-05-05

CONDITIONS: Lyme Disease
Keywords: Lyme Disease; Ixodes scapularis; Borrelia Burgdorferi; Post treatment; Tick bite
MeSH Terms: conditions — Lyme Disease; Tick Bites | interventions — Blood Specimen Collection; Xenodiagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (5):
- Cohort #1: Patients with Lyme disease, post-therapy (Active Comparator): Participants with Lyme disease, post-therapy had 25-30 clean laboratory-reared larval ticks applied as close as possible to the previous site of Lyme disease manifestation. Ticks were secured under a retention dressing and allowed to attach to the research participant. Ticks were removed 3 - 6 days after the placement.
  Interventions: Procedure: Skin biopsy; Procedure: Blood draw; Device: Xenodiagnosis
- Cohort #2: Patients with post-Lyme disease symptoms (PTLDs) (Active Comparator): Participants with post-treatment Lyme disease symptoms (PTLDS) at least 12-months from initial treatment had 25-30 clean laboratory-reared larval ticks applied as close as possible to the previous site of Lyme disease manifestation. Ticks were secured under a retention dressing and allowed to attach to the research participant. Ticks were removed 3 - 6 days after the placement.
  Interventions: Procedure: Skin biopsy; Procedure: Blood draw; Device: Xenodiagnosis
- Cohort #3: New Acute Erythema Migrans (Active Comparator): Participant with new onset of acute erythema migrans had 25-30 clean laboratory-reared larval ticks applied as close as possible to the site of Lyme disease manifestation. Ticks were secured under a retention dressing and allowed to attach to the research participant. Ticks were removed 3 - 6 days after the placement.
  Acute erythema migrans participant (possible positive control)
  Interventions: Procedure: Skin biopsy; Procedure: Blood draw; Device: Xenodiagnosis
- Cohort #4: Untreated Lyme Arthritis (Active Comparator): Participant with untreated Lyme arthritis had 25-30 clean laboratory-reared larval ticks applied as close as possible to the site of Lyme disease manifestation. Ticks were secured under a retention dressing and allowed to attach to the research participant. Ticks were removed 3 - 6 days after the placement.
  Lyme Arthritis participant (possible positive control)
  Interventions: Procedure: Skin biopsy; Procedure: Blood draw; Device: Xenodiagnosis
- Cohort #5: Healthy Volunteers (Active Comparator): Healthy volunteers with no history of Lyme disease had 25-30 clean laboratory-reared larval ticks applied to a body site that was comfortable for participant. Ticks were secured under a retention dressing and allowed to attach to the research participant. Ticks were removed 3 - 6 days after the placement.
  Healthy Volunteers (negative control)
  Interventions: Procedure: Skin biopsy; Procedure: Blood draw; Device: Xenodiagnosis

INTERVENTIONS:
Procedure: Skin biopsy — Optional 2-3mm skin punch biopsies will be performed.
Procedure: Blood draw — Peripheral blood draws will be performed.
Device: Xenodiagnosis — Larval ticks will be obtained from Dr. Sam Telford from a laboratory maintained tick colony at Tufts Veterinary School. These ticks are hatched from eggs laid by ticks that have fed only on specific pathogen free laboratory animals that were purchased from established vendors. Between 25-30 larval ticks that have been aged and are known to be ready to attach will be placed on the study participant.

SUMMARY:
Background:

The most common tick-borne illness in the United States, Lyme disease is caused by Borrelia burgdorferi bacteria that are transmitted to people by Ixodes scapularis ticks. Most cases of Lyme disease are cured by antibiotics, but some patients continue to experience symptoms despite the absence of detectable Lyme bacteria. Xenodiagnosis uses a vector to detect the presence of a disease-causing microbe. Researchers will use live, laboratory-bred ticks to see if Lyme disease bacteria can be detected in people after completing antibiotic therapy and if that is more common in people who continue to experience symptoms such as fatigue and joint pain.

Objectives:

- To see if ticks can be used to detect B. burgdorferi in people who have had Lyme disease and received antibiotic therapy and if it correlates with persistent symptoms.

Eligibility:

* Adults at least 18 years old who have:
* Untreated erythema migrans (the Lyme disease rash); OR
* Untreated Lyme arthritis; OR
* Continuing symptoms after treatment for Lyme disease; OR
* Had Lyme disease and antibiotic treatment within the past 12 months.
* Healthy volunteers

Design:

* Participants will be screened with medical history, physical exam, and blood tests.
* Visit 1:
* Blood and urine tests, health questionnaire.
* Up to 30 laboratory-bred, pathogen-free, larval ticks (each smaller than a poppy seed) will be placed under a dressing.
* Participants may have two small biopsies of skin .
* 4 6 days later, Visit 2:
* Dressing will be removed and ticks will be collected.
* Participants will answer symptom questions.
* If many ticks are still attached, participants will have to come back the next day. If not enough ticks feed successfully, the procedure may be repeated.
* Participants will keep a diary of symptoms for 30 days. Over 3 months, they will be return to the clinic 3 times to see how they feel and answer questionnaires. Test results will be discussed.

DETAILED DESCRIPTION:
Lyme disease is the most common vector borne disease in the United States. Although antibiotic therapy is clinically effective in treating the symptoms of Lyme disease for most patients early in the course of disease, a significant number of patients who receive therapy report persistent symptoms. The cause of persistent symptoms after antibiotic therapy for Lyme disease is an area of great controversy. Recent studies have shown that the organism (Borrelia burgdorferi) may persist in animals after antibiotic therapy and can be detected by using the natural tick vector (Ixodes scapularis) to acquire the organism through feeding (xenodiagnosis). Whether this occurs in humans is unknown. Currently available tests for human Lyme disease do not allow determination of persistent infection after antibiotic therapy.

We performed the first study of the use of I. scapularis larva for the xenodiagnosis of B. burgdorferi infection in humans. Our pilot study showed that xenodiagnosis was well tolerated with no severe adverse events (AEs). The most common AE was mild itching at the site. In this small pilot study, xenodiagnosis for B. burgdorferi was positive in 2 participants and indeterminate in 2 participants. Further studies are needed to determine the sensitivity of xenodiagnosis in evaluating the infection status of Lyme disease patients.

In this proposal, we want to further investigate the utility of xenodiagnosis for identifying persistence of infection with B. burgdorferi in treated human Lyme disease. Our objectives include assessing the link between detection of B. burgdorferi by xenodiagnosis and persistence of symptoms in patients diagnosed with Lyme disease, within 1 year, post therapy; compare the rate of detection of B. burgdorferi by xenodiagnosis after therapy in participants with posttreatment Lyme disease symptoms; identify subject characteristics related to the likelihood of detecting B. burgdorferi by xenodiagnosis including: time from infection, time between infection and therapy, time from therapy; and continue to assess the safety of xenodiagnosis in humans.

The results of study have the potential to resolve this long-standing controversy in Lyme disease pathogenesis. While xenodiagnosis is unlikely to be widely used in clinical practice due to the labor intensity and speed of testing, if our study shows a linkage between positive xenodiagnostic testing and persistence of symptoms after B. burgdorferi infection, it may prove to be a useful tool for testing new strategies for treatment and for correlation with more generally applicable diagnostic markers. Understanding the pathogenesis of persistent symptoms following Lyme disease, and identifying reliable diagnostic tests for determining the success of antibiotic therapy, is critical to the medical management of these patients.

ELIGIBILITY:
* INCLUSION CRITERIA

Criteria for the diagnosis and therapy for Lyme disease can be found at the clinical assessment, treatment, and prevention of Lyme disease, human granulocytic anaplasmosis, and babesiosis: clinical practice guidelines by the Infectious Diseases Society of America.

PATIENTS WITH LYME DISEASE, POST-THERAPY (N=100)

1. Age 18 or older
2. Lyme disease diagnosed in the previous 13 months, fulfilling the case definition of confirmed or probable Lyme disease by the US Centers for Disease Control and Prevention (CDC) (https://wwwn.cdc.gov/nndss/conditions/lyme-disease/case-definition/2017/).
3. Completion of 1 course of antibiotics at least 3 months and up to 12 months between the end of the therapy and the xenodiagnostic procedure.
4. Antibiotic treatment fulfills the Infectious Diseases Society of America guidelines for the recommended therapy for Lyme disease

PATIENTS WITH POST-LYME DISEASE COMPLAINTS AT LEAST 12 MONTHS FROM INITIAL TREATMENT (N=40)

1. Age 18 or older.
2. Diagnosed with confirmed or probable Lyme disease fulfilling the case definition of Lyme disease by the CDC (https://wwwn.cdc.gov/nndss/conditions/lyme-disease/case-definition/2017/).
3. Received recommended antibiotic therapy for Lyme disease 5 at least 12 months between the end of the initial antibiotic therapy and the xenodiagnostic procedure.
4. Persistent or recurrent symptoms that began or worsened within 6 months of the diagnosis and treatment for Lyme disease.

ACUTE EM (N=40)

1. Age 18 or older.
2. EM diagnosed by the study physician.
3. Receiving antibiotic therapy for Lyme disease for less than 48 hours.

LYME ARTHRITIS (N=40)

1. Age 18 or older.
2. Lyme arthritis and have not received antibiotic therapy for the disease.

HEALTHY VOLUNTEERS (N=20)

1. Age 18 or older.
2. No prior history of Lyme disease.
3. Negative whole cell enzyme-linked immunosorbent assay (ELISA) or C6-based antibody test for Lyme disease.

Patients with recently diagnosed (acute) EM (within 48 hours of starting antibiotic therapy) and patients with untreated Lyme arthritis will be recruited in an attempt to increase the chances of finding a positive result by xenodiagnosis (an attempt of a positive control) While patients with acute untreated EM would be the best positive control group, it would be unethical to withhold therapy in these patients for the few days required for tick feeding, due to the risk of dissemination of the organism and possible morbidity. Patients with untreated Lyme arthritis will be recruited to establish whether xenodiagnosis can be used to identify infection in late stage Lyme patients where the bacterium is known to be present. These patients have been infected for months and will not be harmed for delaying therapy for a few days. Lyme arthritis is a late manifestation of B. burgdorferi infection, and hematogenous dissemination already occurred at this late stage. Studies have shown that the presence or absence of previous antibiotic treatment is more predictive than the duration of untreated arthritis for the success of antibiotic therapy in Lyme arthritis. Similarly, patients who just started therapy for EM may still have live Borrelia in the skin and xenodiagnosis may be able to recover the bacteria (but culture of skin biopsies from patients with EM become negative very quickly - within one dose - on antibiotic therapy).

While treatment for Lyme disease will not be offered under this protocol, it may be available via different clinical research protocols or regular medical care at the study site. If not, treatment will be prescribed by the patient's primary care. For patients with untreated early Lyme disease (erythema migrans), antibiotics can be started at the same day of tick placement. For patients with untreated Lyme arthritis, antibiotics can be started after collection of xenodiagnostic ticks (usually 4-5 days, up to 7 days). For patients with Lyme arthritis, if less than 14 ticks fed successfully and if the participant agrees, antibiotic treatment can be delayed until after the repeat procedure.

Patients with acute EM and untreated Lyme arthritis will be able to re-enroll as Patients with Lyme disease, post-therapy. Therefore, in case of positive results, we will be able to compare between the procedures.

Negative control patients will include healthy volunteers from Lyme endemic areas who have never been diagnosed with Lyme disease and have a negative B. burgdorferi ELISA and C6 antibody titer.

EXCLUSION CRITERIA

1. No antibiotic therapy active against Lyme disease in the previous 3 months (except patients with acute EM). Prophylaxis with a single dose of doxycycline 200 mg is not an exclusion.
2. History of allergy to surgical tape or dressing.
3. History of severe reactions to tick bites (granuloma or systemic reactions).
4. Inability to maintain the dressing for any reason.
5. Pregnancy or lactation.
6. Unwillingness to use an effective method of birth control for the duration of participation in the study (women of child-bearing potential only) and for at least 3 months following the last tick placement.
7. Use of investigational therapy and devices during the time of the study and/or in the month prior to signing the informed consent.
8. Active severe skin disease, uncontrolled diabetes, cancer other than non-melanoma skin cancers, autoimmune disease requiring immunosuppressive therapy, or history of HIV, chronic viral hepatitis, or syphilis.
9. Oral or IV steroids in the previous 2 weeks (topical, nasal, inhaled, intra-articular, and replacement doses of steroids are not exclusions).
10. Any other condition that, in the opinion of the investigator, would make the patient unsuitable for enrollment or could interfere with the patient participating in and completing the study.
11. Refusal to participate in specimen collection and storage for future study related use.

EXCLUSION FROM SKIN BIOPSY PART OF THE PROTOCOL

1. History of forming large thick scars (keloids) after skin injuries or surgery.
2. History of excessive bleeding after cuts or procedures.
3. Currently taking anticoagulants.
4. History of allergy to lidocaine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2015-07-24 (Actual); Primary Completion 2022-05-04 (Actual); Study Completion 2022-05-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R Marques, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (5):
- United States (5):
  - Mansfield Family Practice, Storrs, Connecticut
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Tufts Medical Center, Boston, Massachusetts
  - Stony Brook University (State University of New York), Stony Brook, New York
  - New York Medical College, Valhalla, New York

REFERENCES:
- [Background] Marques A, Telford SR 3rd, Turk SP, Chung E, Williams C, Dardick K, Krause PJ, Brandeburg C, Crowder CD, Carolan HE, Eshoo MW, Shaw PA, Hu LT. Xenodiagnosis to detect Borrelia burgdorferi infection: a first-in-human study. Clin Infect Dis. 2014 Apr;58(7):937-45. doi: 10.1093/cid/cit939. Epub 2014 Feb 11. PMID 24523212
- [Background] Telford SR 3rd, Hu LT, Marques A. Is there a place for xenodiagnosis in the clinic? Expert Rev Anti Infect Ther. 2014 Nov;12(11):1307-10. doi: 10.1586/14787210.2014.966084. PMID 25301228
- [Background] Hodzic E, Imai D, Feng S, Barthold SW. Resurgence of persisting non-cultivable Borrelia burgdorferi following antibiotic treatment in mice. PLoS One. 2014 Jan 23;9(1):e86907. doi: 10.1371/journal.pone.0086907. eCollection 2014. PMID 24466286
- [Result] Turk SP, Lumbard K, Liepshutz K, Williams C, Hu L, Dardick K, Wormser GP, Norville J, Scavarda C, McKenna D, Follmann D, Marques A. Post-treatment Lyme disease symptoms score: Developing a new tool for research. PLoS One. 2019 Nov 11;14(11):e0225012. doi: 10.1371/journal.pone.0225012. eCollection 2019. PMID 31710647
- [Derived] Marques AR, Ng SP, McCarthy JE, Telford SR 3rd, Dardick K, Wormser GP, Marcos LA, Tokarz R, Williams C, Law M, Norville J, Lundt M, Petnicki-Ocwieja T, Scavarda C, McKenna D, Goethert HK, Mateja A, Follman D, Eshoo MW, Hu LT. Xenodiagnosis to search for Borrelia burgdorferi after antibiotic treatment of Lyme disease: a prospective cohort study. Clin Infect Dis. 2026 Jan 21:ciag031. doi: 10.1093/cid/ciag031. Online ahead of print. PMID 41563326
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-I-0131.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 72 participants consented, one participant was screen failure and 71 participants started the study.
Groups:
- Cohort #2: Patients With Post-treatment Lyme Disease Symptoms (PTLDs): Participants with post-treatment Lyme disease symptoms (PTLDS) at least 12-months from initial treatment had 25-30 clean laboratory-reared larval ticks applied as close as possible to the previous site of Lyme disease manifestation. Ticks were secured under a retention dressing and allowed to attach to the research participant. Ticks were removed 3 - 6 days after the placement.
Period: Overall Study
Arm/Group | Cohort #1: Patients With Lyme Disease, Post-therapy | Cohort #2: Patients With Post-treatment Lyme Disease Symptoms (PTLDs) | Cohort #3: New Acute Erythema Migrans | Cohort #4: Untreated Lyme Arthritis | Cohort #5: Healthy Volunteers
Started | 40 | 20 | 1 | 1 | 9
Completed | 40 | 20 | 1 | 1 | 9
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort #1: Patients With Lyme Disease, Post-therapy | Cohort #2: Patients With Post-treatment Lyme Disease Symptoms (PTLDs) | Cohort #3: New Acute Erythema Migrans | Cohort #4: Untreated Lyme Arthritis | Cohort #5: Healthy Volunteers | Total
Number analyzed (Participants) | 40 | 20 | 1 | 1 | 9 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 33 | 13 | 1 | 1 | 9 | 57
  >=65 years | 7 | 7 | 0 | 0 | 0 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 9 | 1 | 0 | 4 | 31
  Male | 23 | 11 | 0 | 1 | 5 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 0 | 3 | 5
  Not Hispanic or Latino | 37 | 20 | 1 | 1 | 6 | 65
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 39 | 20 | 1 | 1 | 7 | 68
  More than one race | 1 | 0 | 0 | 0 | 2 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Detection of Borrelia Burgdorferi in Ticks After Xenodiagnosis Procedure
Description: Recovered ticks after feeding on research participants were tested for presence of B. burgdorferi using at least one of three procedures:
  1. Test ticks by polymerase chain reaction (PCR) and culture - Injection of tick lysate into severe combined immunodeficiency (SCID) mice with subsequent PCR and culture testing
  2. Test ticks using isothermal amplification reaction included in the PCR electrospray ionization mass spectroscopy
  3. Test ticks by PCR using the Tick-borne disease Capture Sequencing Assay (TBDCapSeq)
Time Frame: 3-6 days post tick placement
Population: Participants in cohorts 1 & 2 as pre-specified in the protocol.
Measure: Count of Units; unit: Ticks
Units Other Than Participants: Ticks
Arm/Group | Cohort #1: Patients With Lyme Disease, Post-therapy | Cohort #2: Patients With Post-treatment Lyme Disease Symptoms (PTLDs)
Number analyzed (Participants) | 40 | 20
Number analyzed (Ticks) | 419 | 319
Ticks
  Positive | 1 | 0
  Negative | 418 | 319

2. Primary Outcome: Participants With Adverse Event Related to the Application of Ticks (Xenodiagnosis)
Description: Safety of xenodiagnosis in humans was assessed by number of participants with adverse event related to the application of ticks. Adverse event was assessed using participants self-reported diary cards and clinical interview.
Time Frame: Up to 30-days after tick removal
Population: All participants in who started the study
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort #1: Patients With Lyme Disease, Post-therapy | Cohort #2: Patients With Post-treatment Lyme Disease Symptoms (PTLDs) | Cohort #3: New Acute Erythema Migrans | Cohort #4: Untreated Lyme Arthritis | Cohort #5: Healthy Volunteers
Number analyzed (Participants) | 40 | 20 | 1 | 1 | 9
Participants
  Application site itching | 24 | 13 | 0 | 1 | 5
  Other application site reaction | 13 | 8 | 0 | 1 | 3

ADVERSE EVENTS:
Time Frame: Up to 30 days post tick removal
Arm/Group | Cohort #1: Patients With Lyme Disease, Post-therapy | Cohort #2: Patients With Post-treatment Lyme Disease Symptoms (PTLDs) | Cohort #3: New Acute Erythema Migrans | Cohort #4: Untreated Lyme Arthritis | Cohort #5: Healthy Volunteers
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/20 | 0/1 | 0/1 | 0/9
Serious Adverse Events (participants affected / at risk) | 1/40 | 3/20 | 0/1 | 0/1 | 0/9
Other Adverse Events (participants affected / at risk) | 35/40 | 19/20 | 1/1 | 1/1 | 6/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort #1: Patients With Lyme Disease, Post-therapy (N=40) | Cohort #2: Patients With Post-treatment Lyme Disease Symptoms (PTLDs) (N=20) | Cohort #3: New Acute Erythema Migrans (N=1) | Cohort #4: Untreated Lyme Arthritis (N=1) | Cohort #5: Healthy Volunteers (N=9)
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort #1: Patients With Lyme Disease, Post-therapy (N=40) | Cohort #2: Patients With Post-treatment Lyme Disease Symptoms (PTLDs) (N=20) | Cohort #3: New Acute Erythema Migrans (N=1) | Cohort #4: Untreated Lyme Arthritis (N=1) | Cohort #5: Healthy Volunteers (N=9)
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0 | 0 | 0
Photophobia (Eye disorders) | 1 | 0 | 0 | 0 | 0
Uveitis (Eye disorders) | 1 | 0 | 0 | 0 | 0
Visual disturbance NOS (Eye disorders) | 1 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 4 | 0 | 0 | 0
Gastroenteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 2 | 0 | 0 | 1
Pyrosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Application Site Discharge (General disorders) | 0 | 1 | 0 | 0 | 0
Application site erythema (General disorders) | 2 | 0 | 0 | 0 | 0
Application site pain (General disorders) | 8 | 2 | 0 | 0 | 2
Application Site Papule (General disorders) | 1 | 1 | 0 | 0 | 0
Application site pruritus (General disorders) | 24 | 13 | 0 | 1 | 5
Application site redness (General disorders) | 1 | 0 | 0 | 0 | 1
Application site swelling (General disorders) | 1 | 0 | 0 | 0 | 0
Application site tenderness (General disorders) | 5 | 6 | 0 | 1 | 1
Application site vesicles (General disorders) | 0 | 2 | 0 | 0 | 1
Fatigue (General disorders) | 4 | 2 | 0 | 1 | 0
Fever (General disorders) | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 1
Thirst (General disorders) | 1 | 1 | 0 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 0
Injury (Injury, poisoning and procedural complications) | 2 | 1 | 0 | 0 | 0
Insect bite NOS (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 3 | 0 | 0 | 2
Muscle ache (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 3 | 0 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Neck stiffness (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0 | 0
Cognitive function abnormal (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 12 | 4 | 1 | 0 | 4
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Sleep disturbances (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Mood alteration NOS (Psychiatric disorders) | 2 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2
Surgery (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-22): https://cdn.clinicaltrials.gov/large-docs/26/NCT02446626/Prot_SAP_000.pdf